CLINICAL TRIAL: NCT01216488
Title: Comparison of Axillary Block Under Ultrasound With 40 or 25 ml of Xylocaine 1.5% Adrenalin in Forearm or Arm Surgery.
Brief Title: Comparison Between Two Different Volumes of Anesthesia Drug in Forearm Surgery
Acronym: COMBAX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RB09-060
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2011-12-21 (Estimated); Status verified 2011-12

CONDITIONS: Forearm and Arm Surgery
Keywords: Forearm surgery; Hand surgery; Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 40 ml of Xylocaine (Active Comparator)
  Interventions: Drug: Xylocaine
- 25 ml of Xylocaine (Experimental)
  Interventions: Drug: Xylocaine

INTERVENTIONS:
Drug: Xylocaine — 40 ml or 25 ml of Xylocaine injection

SUMMARY:
Hospitalized patients for superior member surgery have different types of anesthesia.Forearm and/or arm surgery could be done under general anesthesia, but in the most of the cases, this surgery was done under locoregional anesthesia.Several injections of local anesthesia at the nerves axilla are used with the used of ultrasonography.

The purpose of this study is to show that the anesthesia efficiency is the same with 40 or 25 ml of Xylocaine 1.5% Adrenalin in Forearm or Arm Surgery.

DETAILED DESCRIPTION:
Inclusion criteria :

* age > 18 years old
* patient who must have a non emergency surgery of the forearm or the hand
* ASA I or ASA II
* informed consent
* Ensured patient

Exclusion criteria :

* pregnancy
* respiratory insufficiency
* cardiac insufficiency
* hepatic insufficiency
* renal insufficiency
* ASA III or IV
* contraindications to the locoregional anesthesia
* contraindications to the xylocaine used
* patient participate to an another clinical study
* guardianship patient

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* patient who must have a non emergency surgery of the forearm or the hand
* ASA I or ASA II
* informed consent
* Ensured patient

Exclusion Criteria:

* pregnancy
* respiratory insufficiency
* cardiac insufficiency
* hepatic insufficiency
* renal insufficiency
* ASA III or IV
* contraindications to the locoregional anesthesia
* contraindications to the xylocaine used
* patient participate to an another clinical study
* guardianship patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Axillary block efficiency conducted by ultrasound | 48 hours
  during the hospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: François PICART, MD, Principal Investigator — CHRU Brest
Locations (1):
- Department of Anesthesia CHRU Brest, Brest, Brittany Region, France